CLINICAL TRIAL: NCT02200354
Title: The Safety and Efficacy of Pemetrexed Rechallenge With Bevacizumab for Patients With Advanced Non-squamous Non-small Cell Lung Cancer
Brief Title: The Safety and Efficacy of Pemetrexed Rechallenge With Bevacizumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inclusion speed
Sponsor: Kobe City General Hospital (Other)
Responsible Party: Principal Investigator, Daichi Fujimoto, doctor, division of respiratory medicine, Kobe City General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEM-RE-2014
Record Dates: First submitted 2014-07-20; First posted 2014-07-25 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — Pemetrexed; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pemetrexed with bevacizumab (Experimental): pemetrexed rechallenge with bevacizumab pemetrexed (500mg/m2 day1) bevacizumab (15mg/kg day1)
  Interventions: Drug: pemetrexed with bevacizumab

INTERVENTIONS:
Drug: pemetrexed with bevacizumab

SUMMARY:
For patients with nonsquamous NSCLC and a good performance status (PS), pemetrexed and cisplatin has been recommended for first-line NSCLC treatment. Recently, results from the PARAMOUNT trial showed that patients with nonsquamous NSCLC who had a good PS and had not progressed after completing four cycles of pemetrexed-cisplatin induction therapy benefitted from pemetrexed continuation maintenance therapy. Furthermore, pemetrexed with bevacizumab continuous maintenance might be better treatment option, considering the results from AVAPEARL trial. Pemetrexed rechallenge has been reported to be effective in some patients. Therefore, in order to investigate the safety and efficacy of pemetrexed rechallenge with bevacizumab,we conducted this study.

ELIGIBILITY:
Inclusion Criteria:

* 20 Years and older
* PS0-2
* Advanced non-squamous non-small cell lung cancer; AND
* Patients who have received more than 4 cycles of pemetrexed therapy before the study

Exclusion Criteria:

* Interstitial pneumonia; AND
* Abnormal blood test

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2018-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
progression free survival | Within the study period and until tumor proression, an expected average of 16 weeks

SECONDARY OUTCOMES:
response rate | The response will be assessed while participants received the pemetrexed with bevacizumab, an expected average to the maximum response of 4 - 16 weeks
overall survival | From date of the start of pemetrexed with bevacizumab until date of death from any cause, up to 3 years
time to treatment failure (TTF) | From date of the start of pemetrexed with bevacizumab until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
Number of Participants with Adverse Events | From date of the start of pemetrexed with bevacizumab until the participants stop this therapy, an expected average of 16 weeks and up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daichi Fujimoto, MD, Principal Investigator — Kobe City Medical Center General Hospital
Locations (1):
- Kobe City Medical Center General Hospital, Kobe, Hyōgo, Japan